CLINICAL TRIAL: NCT05516251
Title: Transcutaneous Supraorbital Nerve Stimulator Versus Topiramate in Prevention of Recurrent Migraine: A Prospective, Randomized Comparative Study.
Brief Title: Transcutaneous Supraorbital Nerve Stimulator Versus Topiramate in Prevention of Recurrent Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-S203
Record Dates: First submitted 2022-08-16; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Migraine, Classic
MeSH Terms: conditions — Migraine with Aura | interventions — Topiramate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topiramate (Active Comparator)
  Interventions: Drug: Topiramate 25Mg Tab
- Transcutaneous Supraorbital Nerve Stimulator (Experimental)
  Interventions: Device: Transcutaneous Supraorbital Nerve Stimulator

INTERVENTIONS:
Device: Transcutaneous Supraorbital Nerve Stimulator — SNS devices (DJTT-Ib, Hengyang Dajing Medical Instrument Technology Co., Ltd.) Stimulation electrodes are placed on the bilateral forehead, covering the supratrochlear and supraorbital nerves. The stimulus parameters are set as follows: pulse width 300 μsec, frequency 60 Hz, pulse duration μsec, increasing current peaked at 14 min with 16 mA. Patients receive SNS treatment daily for 20 min, no lease than 5 per week, last for 4 weeks.
  Arms: Transcutaneous Supraorbital Nerve Stimulator
Drug: Topiramate 25Mg Tab — Topiramate 25Mg Tab (Tuotai Pian, Xian Janssen Pharmaceutical Ltd.) are prescribed to participates by one neurologist. Participates are asked to take 25mg oral per day in a fixed time usually in the morning.
  Arms: Topiramate

SUMMARY:
Migraine has been ranked as the second most disabling neurological disorder in the worldwide. Medication or nonpharmacological treatments are all reasonable options for the prevention. Oral topiramate treatment is a typical effective method, while transcutaneous supraorbital nerve stimulation (SNS) was reported to be valuable for migraine acute treatment and even the prevention. As a new nonpharmacological therapeutic method, whether SNS is equivalent to topiramate is still unknown. The aim of the present study was to compare their effects in a cohort of migraine patients. After diagnosed with recurrent or chronic migraine and consented to this research, patients received randomly treatments by either SNS or topiramate, and were followed up prospectively. After a 1-month period of baseline observation, patients were followed by a 1-month treatment, and next 2-month period of followup. At least the following assessments will be performed: (1) Change from baseline in the number of migraine days during the 3 observing months; (2) Change from baseline in the number of moderate/ severe headache days over the 3 observing months; (3) 50% responder rate for the reduction of migraine days (percentage of patients having at least 50% reduction of migraine days) during the first treating month. Comparison of outcome measures between the 2 treatment groups will be performed to show the equivalence of SNS versus topiramate.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-60 years old;
* Diagnosed with definite migraine (ICHD-3 code 1.1 or 1.2);
* At least 2 migraine attacks per month during the past 3 months;
* Consent to participate in the study;
* No contraindications to associated treatments.

Exclusion Criteria:

* Received preventive treatments during the previous 3 months;
* Definite other kinds of headache, especially tension-type, medication overuse and secondary headache (ICHD-3 code 8.2);
* Severe neurological or psychiatric disorders;
* Severe primary systemic disorders including heart, brain, liver, kidney, and hematopoietic system;
* Women with pregnancy or lactation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
migraine days | during the 3 observing months
  Change from baseline in the number of migraine days during the 3 observing months
moderate/ severe headache days | over the 3 observing months
  Change from baseline in the number of moderate/ severe headache days over the 3 observing months
50% responder rate | during the first treating 1 month
  50% responder rate for the reduction of migraine days (percentage of patients having at least 50% reduction of migraine days) during the first treating month

SECONDARY OUTCOMES:
Averaged migraine days | during the 3 observing months
  Averaged migraine days per 4 weeks
migraine attacks | during the 3 observing months
  Number of migraine attacks per 4 weeks
Cumulative pain hours | during the 3 observing months
  Cumulative hours per 4 weeks of moderate/severe pain (Suggested by visual analogue scale)
bothersome symptoms | during the 3 observing months
  Effect on the most bothersome symptoms (anorexia, nausea, vomiting, photophobia, phonophobia. Weakness and dizziness)
Migraine functional impact | during the 3 observing months
  Using Headache Impact Test-6 (HIT-6) questionnaire, migraine functional impact were evaluated per 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyuan Yu, Study Director — Tongji Hospital
Locations (1):
- Wensheng Qu, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Riederer F, Penning S, Schoenen J. Transcutaneous Supraorbital Nerve Stimulation (t-SNS) with the Cefaly(R) Device for Migraine Prevention: A Review of the Available Data. Pain Ther. 2015 Oct 14;4(2):135-47. doi: 10.1007/s40122-015-0039-5. Online ahead of print. PMID 26467451
- [Result] Ordas CM, Cuadrado ML, Pareja JA, de-Las-Casas-Camara G, Gomez-Vicente L, Torres-Gaona G, Venegas-Perez B, Alvarez-Marino B, Diez Barrio A, Pardo-Moreno J. Transcutaneous Supraorbital Stimulation as a Preventive Treatment for Chronic Migraine: A Prospective, Open-Label Study. Pain Med. 2020 Feb 1;21(2):415-422. doi: 10.1093/pm/pnz119. PMID 31131857
- [Result] Vikelis M, Dermitzakis EV, Spingos KC, Vasiliadis GG, Vlachos GS, Kararizou E. Clinical experience with transcutaneous supraorbital nerve stimulation in patients with refractory migraine or with migraine and intolerance to topiramate: a prospective exploratory clinical study. BMC Neurol. 2017 May 18;17(1):97. doi: 10.1186/s12883-017-0869-3. PMID 28521762